CLINICAL TRIAL: NCT01502293
Title: A Multicenter Phase II Trial of Intratumoral pIL-12 Electroporation in Advanced Stage Cutaneous and in Transit Malignant Melanoma
Brief Title: Trial of pIL-12 Electroporation Malignant Melanoma
Acronym: IL-12MEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OncoSec Medical Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMS-I100; 11854 (Other: University of California, San Francisco)
Record Dates: First submitted 2011-12-21; First posted 2011-12-30 (Estimated); Results first posted 2019-09-26 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Main Study: tavo-EP (Experimental): Patients received one cycle (3 daily treatments on Days 1, 5, and 8) of intra-tumoral injection(s) of tavo at a fixed dose of 0.5 mg/mL (up to 4 tumor sites) followed immediately by in vivo electroporation. Treatment could be repeated at 3-month intervals until disease progression or unacceptable toxicity for up to 5 cycles.
  Interventions: Biological: Tavokinogene Telseplasmid (tavo); Device: OncoSec Medical System (OMS)
- Addendum: Regimen A tavo-EP (Experimental): Patients received one cycle (3 daily treatments on Days 1, 8, and 15) of intra-tumoral injection(s) of tavo at a fixed dose of 0.5 mg/mL (up to 4 tumor sites) followed immediately by in vivo electroporation. Treatment could be repeated at 6-week intervals until disease progression or unacceptable toxicity for up to 9 cycles.
  Interventions: Biological: Tavokinogene Telseplasmid (tavo); Device: OncoSec Medical System (OMS)
- Addendum: Regimen B tavo EP (Experimental): Patients received one cycle (3 daily treatments on Days 1, 5, and 8) of intra-tumoral injection(s) of tavo at a fixed dose of 0.5 mg/mL (up to 4 tumor sites) followed immediately by in vivo electroporation. Treatment could be repeated at 6-week intervals until disease progression or unacceptable toxicity for up to 2 cycles.
  Interventions: Biological: Tavokinogene Telseplasmid (tavo); Device: OncoSec Medical System (OMS)

INTERVENTIONS:
Biological: Tavokinogene Telseplasmid (tavo) — Patients received intratumoral injection(s) of tavo.
  Other Names: interleukin-12 gene; IL-12 gene; pIL-12; plasmid DNA encoding human interleukin-12; plasmid IL-12 Device: OncoSec Med
Device: OncoSec Medical System (OMS) — Electroporation via OMS was performed immediately following intratumoral injection of tavo. A sterile applicator containing 6 stainless steel electrodes arranged in a circle were placed around the tumor. The applicator was connected to the OMS power supply and six pulses were administered to each tumor lesion at the approximate point of tavo injection.
  Other Names: MedPulser

SUMMARY:
This study will assess the safety and effectiveness of different dosing regimens of ImmunoPulse IL-12® in malignant melanoma. ImmunoPulse IL-12® is the combination of intratumoral interleukin-12 gene (also known as tavokinogene telseplasmid [tavo]) and in vivo electroporation-mediated plasmid deoxyribonucleic acid [DNA] vaccine therapy (tavo-EP) administered using the OncoSec Medical System (OMS). ImmunoPulse IL-12® is a gene therapy approach to directly induce a pro-inflammatory response within a tumor to initiate and/or enhance anti-tumor immunity.

DETAILED DESCRIPTION:
Plasmid IL-12 (pIL-12) at a concentration of 0.5 mg/mL will be injected intratumorally at a dose volume of ¼ of the calculated lesion volume and a dose volume per lesion of 0.1 mL for lesions of volume < 0.4 cm3. Six pulses at field strengths of (E+) of 1500 V/cm and pulse width of 100 μs at 1-second intervals will be administered using the OncoSec Medical System (OMS) to each previously injected tumor.

Three treatment regimens will be explored:

Main Study: Treatment on Days 1, 5 and 8 for 1 cycle. Additional cycles may be repeated every 3 months at the Investigator's discretion.

Addendum Regimen A: Treatment on Days 1, 8 and 15 every 6 weeks. Subsequent cycles may be given at 6-week intervals, for up to 9 treatment cycles in total.

Addendum Regimen B: Treatment on Days 1, 5 and 8 every 6 weeks. Subsequent cycles may be given at 6-week intervals, for up to 9 treatment cycles in total.

NOTE: An Addendum was added to the Main Protocol with the purpose of exploring the safety and efficacy of an increased treatment frequency schedule.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced cutaneous or subcutaneous in-transit or metastatic melanoma (main and addendum)
* Age ≥ 18 years of age (main and addendum).
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (main and addendum).
* Patients may have had prior chemotherapy or immunotherapy (vaccines, interferon, ipilimumab, or IL-2) with progression or persistent disease. All chemotherapy or immunotherapy (prior therapies for cancer per the addendum) must have been stopped 4 weeks prior to electroporation (main part) or prior to enrollment (addendum), unless the sponsor medical monitor approval was obtained.
* Patients may have had radiation therapy, but must have progressive disease after radiation therapy if the lesions to be treated are within the radiation field. Per the main study Protocol Amendment 10 (Version 11.0), dated 27 April 2016, all prior treatment toxicities had to be resolved to Grade 1. Per the study Addendum Amendment 5, dated 27 April 2016, all prior chemotherapy or immunotherapy treatment-related adverse events (AEs) must have been resolved to baseline or Grade 1 at the time of study enrollment; and all prior radiation treatment AEs must have been resolved to baseline at the time of study enrollment.
* Had a minimum of 2 eligible tumors and could have had up to 4 eligible tumors treated with electroporation (main part).
* Must have had a lesion at baseline eligible for treatment, meeting all of the following criteria: at least 0.3 cm x 0.3 cm in longest perpendicular diameters; and accessible for electroporation (addendum).
* Must have had at least 1 additional lesion that could have been followed for distant regression and that met all of the following criteria: must have remained untreated for duration of the study; and had longest perpendicular diameters at least 0.3 cm x 0.3 cm by clinical measurement; or at least 1.0 cm x 1.0 cm by computed tomography (CT) for non-nodal lesions; or at least 1.5 cm x 1.5 cm by CT for malignant lymph nodes (addendum).
* For women of childbearing potential, a negative serum or urine pregnancy test within 14 days to the first study drug administration, and use of birth control from 30 days prior to the first day of study drug administration and 30 days following last day study drug administration was required. Male patients must have been surgically sterile, or must have agreed to use contraception during the study and at least 30 days following the last day of study drug administration (addendum).
* Had a creatinine level < 2 x upper limit of normal (ULN), and serum bilirubin within institutional normal limits obtained within 4 weeks prior to enrollment (main part and addendum).
* Had aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 1.5 x ULN within 4 weeks prior to enrollment (addendum).
* Had an absolute neutrophil count (ANC) > 1000/mm and platelet count > 100,000 /mm within 4 weeks prior to registration (main part) or enrollment (addendum).
* Were able to give informed consent and to follow guidelines given in the study (main part and addendum).

Exclusion Criteria:

* Prior therapy with IL-12 or prior gene therapy (main and addendum).
* Had an ECOG performance score of 3 or 4 (main part).
* Concurrent immunotherapy, chemotherapy, or radiation therapy for duration of patient participation on study (main part and addendum). For the study addendum, approved anti PD1 agents could have been permitted at the investigator's discretion and in consultation with the sponsor's medical monitor.
* Evidence of significant active infection (e.g., pneumonia, cellulitis, wound abscess, etc.) at time of study entry (main part) or enrollment (study addendum).
* Pregnant or breast-feeding women (main part and addendum).
* Women of childbearing age must have had a negative pregnancy test and had to be willing to use a highly effective method of contraception. Men who were sexually active must also have been willing to use an accepted and effective method of contraception (main part).
* Patients with electronic pacemakers or defibrillators are excluded from this study (main part and addendum).
* The patient is known to be positive for Human Immunodeficiency Virus (HIV) or has another confirmed or suspected immunosuppressive or immunodeficient condition (patients with thyroiditis are eligible) (addendum).
* Life expectancy of less than 6 months (main part and addendum).
* Had significant disease or uncontrolled disease, ie, cardiovascular renal, hepatic, endocrine, metabolic, neurologic, or other significant disease that could have limited the patient's ability to participate in the study as determined by the investigator or medical monitor (main part).
* History of significant cardiovascular disease (i.e. New York Heart Association (NYHA) class 3 congestive heart failure; myocardial infarction with the past 6 months; unstable angina; coronary angioplasty with the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias) (study addendum).
* Other clinically significant co-morbidities such as uncontrolled pulmonary disease, uncontrolled diabetes, active central nervous system (CNS) disease, active infection or any other condition that could compromise the patients participation in the study according to the investigator (study addendum).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-02-14 (Actual); Primary Completion 2016-03-21 (Actual); Study Completion 2016-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCSF Helen Diller Comprehensive Cancer Center, San Francisco, California
  - John Wayne Cancer Institute, Santa Monica, California
  - University of Colorado Denver, Denver, Colorado
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Seattle Cancer Care Alliance /University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Algazi A, Bhatia S, Agarwala S, Molina M, Lewis K, Faries M, Fong L, Levine LP, Franco M, Oglesby A, Ballesteros-Merino C, Bifulco CB, Fox BA, Bannavong D, Talia R, Browning E, Le MH, Pierce RH, Gargosky S, Tsai KK, Twitty C, Daud AI. Intratumoral delivery of tavokinogene telseplasmid yields systemic immune responses in metastatic melanoma patients. Ann Oncol. 2020 Apr;31(4):532-540. doi: 10.1016/j.annonc.2019.12.008. Epub 2020 Feb 1. PMID 32147213

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 6 investigative sites in the United States from 14 February 2012 to 21 March 2016.
Groups:
- Addendum: Regimen B Tavo-EP: Patients received one cycle (3 daily treatments on Days 1, 5, and 8) of intra-tumoral injection(s) of tavo at a fixed dose of 0.5 mg/mL (up to 4 tumor sites) followed immediately by in vivo electroporation. Treatment could be repeated at 6-week intervals until disease progression or unacceptable toxicity for up to 2 cycles.
Period: Overall Study
Arm/Group | Main Study: Tavo-EP | Addendum: Regimen A Tavo-EP | Addendum: Regimen B Tavo-EP
Started | 30 | 17 | 4
Completed | 5 | 0 | 0
Not Completed | 25 | 17 | 4
Not completed — Progressive Disease | 20 | 12 | 2
Not completed — Withdrawal by Subject | 3 | 3 | 1
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Reason Not Specified | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, all patients who were enrolled and received any amount of the study treatment (pIL-12).
Groups:
- Total: Total of all reporting groups
Arm/Group | Main Study: Tavo-EP | Addendum: Regimen A Tavo-EP | Addendum: Regimen B Tavo-EP | Total
Number analyzed (Participants) | 30 | 17 | 4 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (10.19) | 68.4 (13.47) | 58.8 (3.30) | 66.7 (11.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 4 | 0 | 18
  Male | 16 | 13 | 4 | 33
Region of Enrollment [Number; unit: participants]
  United States | 30 | 17 | 4 | 51

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Objective Response Rate (ORR) by Modified "Skin" RECIST
Description: ORR is defined as the percentage of participants with evaluable lesions that achieved a complete response (CR) or partial response (PR) as assessed by the investigator using Modified "Skin" Response Evaluation Criteria In Solid Tumors (RECIST). CR: complete disappearance of all lesions (whether measurable or not) and the absence of new lesions for at least 4 weeks duration, confirmed by additional scan and visit 4 to 6 weeks after first documentation of CR. PR: ≥30% decrease in longest dimension (LD) from baseline lesion, and no new lesions.
Time Frame: Main Study: Screening and Days 90, 180, 270 and 360; Addendum: Screening and Weeks 12, 24, 36, and 48
Population: Efficacy Analysis Set, all enrolled patients who received at least one full cycle of study treatment and had at least one efficacy assessment following the first dose of study drug, who had at least one post-baseline response assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Main Study: Tavo-EP | Addendum: Regimen A Tavo-EP | Addendum: Regimen B Tavo-EP
Number analyzed (Participants) | 28 | 16 | 4
percentage of participants | 32.1 | 25.0 | 25.0

2. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, medical treatment or procedure and which did not necessarily have to have had a causal relationship with this treatment. An adverse event could have, therefore, been any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, medical treatment or procedure whether or not considered related to the medicinal product. An SAE was defined an any untoward medical occurrence that at any dosage resulted in one or more of the following: death, A life-threatening adverse event (real risk of dying), inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly, required intervention to prevent permanent impairment of damage.
Time Frame: From first administration of study treatment up to 30 days after last dose or until initiation of new anti-cancer treatment.
Population: Safety Analysis Set, all patients who were enrolled and received any amount of the study treatment (pIL-12).
Measure: Number; unit: percentage of participants
Groups:
- Addendum: Regimen B: Patients received one cycle (3 daily treatments on Days 1, 5, and 8) of intra-tumoral injection(s) of tavo at a fixed dose of 0.5 mg/mL (up to 4 tumor sites) followed immediately by in vivo electroporation. Treatment could be repeated at 6-week intervals until disease progression or unacceptable toxicity for up to 2 cycles.
Arm/Group | Main Study: Tavo-EP | Addendum: Regimen A Tavo-EP | Addendum: Regimen B
Number analyzed (Participants) | 30 | 17 | 4
percentage of participants
  AEs | 96.7 | 94.1 | 50.0
  SAEs | 6.7 | 17.6 | 0

3. Secondary Outcome: Median Overall Survival (OS)
Description: Overall survival (OS) time is defined as the duration between the date of treatment initiation (Study Day 1) to the date of death, regardless of the cause of death, assessed up to 30 months.
Time Frame: From the start of study treatment until death, assessed up to 30 months.
Population: Efficacy Analysis Set, all enrolled patients who received at least one full cycle of study treatment and had at least one efficacy assessment following the first dose of study drug. Patients were censored at the last date that they were known to be alive.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Addendum: Regimen A: Patients received one cycle (3 daily treatments on Days 1, 8, and 15) of intra-tumoral injection(s) of tavo at a fixed dose of 0.5 mg/mL (up to 4 tumor sites) followed immediately by in vivo electroporation. Treatment could be repeated at 6-week intervals until disease progression or unacceptable toxicity for up to 9 cycles.
Arm/Group | Main Study: Tavo-EP | Addendum: Regimen A | Addendum: Regimen B Tavo-EP
Number analyzed (Participants) | 28 | 16 | 4
days | NA [NA to NA] — Median not estimable as all participants were alive at the time of their final follow-up. | NA [NA to NA] — Median not estimable as all participants were alive at the time of their final follow-up. | NA [NA to NA] — Median not estimable as all participants were alive at the time of their final follow-up.

4. Secondary Outcome: Objective Response Rate (ORR) by Immune Related Response Criteria (irRC)
Description: ORR is defined as the percentage of participants with evaluable lesions that achieved a complete response (CR) or partial response (PR) as assessed by the investigator using irRC criteria. CR: complete disappearance of all lesions (whether measurable or not) and the absence of new lesions for at least 4 weeks duration, confirmed by additional scan and visit 4 to 6 weeks after first documentation of CR. PR: ≥50% decrease in the product of the diameters from baseline.
Time Frame: Main Study: Screening and Days 90, 180, 270 and 360; Addendum: Screening and Weeks 12, 24, 36, and 48
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Main Study: Tavo-EP | Addendum: Regimen A Tavo-EP | Addendum: Regimen B Tavo-EP
Number analyzed (Participants) | 28 | 16 | 4
percentage of participants | 28.6 | 25.0 | 0

5. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response (CR or PR based on Modified RECIST criteria) is defined as the number of days from the initial documentation of an objective response to the most current evaluation of that response or to documentation of progression or death associated with disease progression. CR: complete disappearance of all lesions (whether measurable or not) and the absence of new lesions for at least 4 weeks duration, confirmed by additional scan and visit 4 to 6 weeks after first documentation of CR. PR: ≥30% decrease in longest dimension (LD) from baseline lesion, and no new lesions. Patients who had an initial response and did not progress were censored at their date of last assessment.
Time Frame: From first documented response until disease progression (Up to 29.7 months)
Population: Efficacy Analysis Set, all enrolled patients who received at least one full cycle of study treatment and had at least one efficacy assessment following the first dose of study drug, who had at least one post-baseline response assessment and had a CR or PR.
Measure: Median (Full Range); unit: days
Arm/Group | Main Study: Tavo-EP | Addendum: Regimen A Tavo-EP | Addendum: Regimen B Tavo-EP
Number analyzed (Participants) | 28 | 16 | 4
days | 96 [22 to 678] | 127 [1 to 169] | NA [NA to NA] — Median not estimable due to low number of participants with objective response.

6. Secondary Outcome: Time to First Objective Response
Description: Time to objective response (CR or PR based on Modified RECIST criteria) is defined as the number of days between the date of treatment initiation (Study Day 1) to the first date of the first documentation of an objective response. CR: complete disappearance of all lesions (whether measurable or not) and the absence of new lesions for at least 4 weeks duration, confirmed by additional scan and visit 4 to 6 weeks after first documentation of CR. PR: ≥30% decrease in longest dimension (LD) from baseline lesion, and no new lesions. Patients who had an initial response and did not progress were censored at their date of last assessment. Patients who did not have an objective response were censored at their date of last assessment.
Time Frame: From start of study treatment until overall objective response (Up to 29.7 months)
Population: as for outcome 5
Measure: Median (Full Range); unit: days
Groups:
- Addendum: Regimen B Tavo-EP: Patients received cycle (3 daily treatments on Days 1, 5, and 8) of intra-tumoral injection(s) of tavo at a fixed dose of 0.5 mg/mL (up to 4 tumor sites) followed immediately by in vivo electroporation. Treatment could be repeated at 6-week intervals until disease progression or unacceptable toxicity for up to 2 cycles.
Arm/Group | Main Study: Tavo-EP | Addendum: Regimen A Tavo-EP | Addendum: Regimen B Tavo-EP
Number analyzed (Participants) | 34 | 16 | 4
days | 88 [38 to 904] | 84 [26 to 381] | 77.5 [69 to 78]

7. Secondary Outcome: Median Progression Free Survival
Description: Progression free survival (PFS) is defined as the duration between the date of treatment initiation (Study Day 1) to the first date of either disease progression at either local or distant sites, or death from any cause. Disease progression at local or distant lesions is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression). Patients were censored at their last assessment date if there was no evidence of disease progression.
Time Frame: From start of study treatment until disease progression or death (Up to 29.7 months)
Population: Efficacy Analysis Set, all enrolled patients who received at least one full cycle of study treatment and had at least one efficacy assessment following the first dose of study drug, who had at least one post-baseline response assessment and had a CR or PR based on Modified RECIST criteria.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Main Study: Tavo-EP | Addendum: Regimen A Tavo-EP | Addendum: Regimen B Tavo-EP
Number analyzed (Participants) | 28 | 16 | 4
days | 96.5 [38 to 762] | 91.5 [6 to 254] | 78 [77 to 107]

8. Secondary Outcome: Regression Rate of Treated and Untreated Lesions
Description: The treated (injected, electroporated) lesion regression rate is defined as the percentage of patients who had at least one treated lesion that decreased in longest dimension by ≥ 30%. The untreated (non-injected, non-electroporated) lesion regression rate is defined as the percentage of patients who had at least one untreated lesion that decreased in longest dimension by ≥ 30%.
Time Frame: Main Study: Screening and Days 1, 39, 90, 120, 180, 270, 360, End Of Study; Addendum: Screening and Weeks 12, 24, 36,28, End of Study
Population: Efficacy Analysis Set, all enrolled patients who received at least one full cycle of study treatment and had at least one efficacy assessment following the first dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Main Study: Tavo-EP | Addendum: Regimen A Tavo-EP | Addendum: Regimen B Tavo-EP
Number analyzed (Participants) | 28 | 16 | 4
percentage of participants
  Treated: number analyzed (Participants) | 25 | 15 | 4
  Treated | 64.0 | 60.0 | 25.0
  Untreated: number analyzed (Participants) | 22 | 13 | 2
  Untreated | 31.8 | 38.5 | 50.0

ADVERSE EVENTS:
Time Frame: From first administration of study treatment up to 30 days after last dose or until initiation of new anti-cancer treatment.
Arm/Group | Main Study: Tavo-EP | Addendum: Regimen A Tavo-EP | Addendum: Regimen B Tavo-EP
Serious Adverse Events (participants affected / at risk) | 2/30 | 3/17 | 0/4
Other Adverse Events (participants affected / at risk) | 29/30 | 16/17 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: Tavo-EP (N=30) | Addendum: Regimen A Tavo-EP (N=17) | Addendum: Regimen B Tavo-EP (N=4)
Cellulitis (Infections and infestations) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Study: Tavo-EP (N=30) | Addendum: Regimen A Tavo-EP (N=17) | Addendum: Regimen B Tavo-EP (N=4)
Eye irritation (Eye disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 5 | 3 | 1
Injection site discolouration (General disorders) | 4 | 2 | 0
Injection site inflammation (General disorders) | 4 | 2 | 0
Chills (General disorders) | 2 | 2 | 0
Oedema peripheral (General disorders) | 2 | 1 | 0
Pyrexia (General disorders) | 2 | 1 | 0
Chest discomfort (General disorders) | 1 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 1
Injection site discharge (General disorders) | 2 | 0 | 0
Injection site erythema (General disorders) | 2 | 0 | 0
Injection site pain (General disorders) | 0 | 2 | 0
Injection site pruritus (General disorders) | 1 | 1 | 0
Pain (General disorders) | 2 | 0 | 0
Injection site laceration (General disorders) | 0 | 1 | 0
Tenderness (General disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 2 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 24 | 12 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 5 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Lymphoedema (Vascular disorders) | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
An Addendum was added to the Main Protocol with the purpose of exploring the safety and efficacy of an increased treatment frequency schedule.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less